CLINICAL TRIAL: NCT02103647
Title: A Randomized, Open-label, Crossover Clinical Trial to Compare The Pharmacokinetics of A Pregabalin Controlled Release Tablet 300mg and Immediate Release Formulation After Multiple Dosing Under Fasted Condition in Healthy Male Subjects
Brief Title: Clinical Trial to Compare The Pharmacokinetics of A Pregabalin Controlled Release Tablet 300mg and Immediate Release Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: IlDong Pharmaceutical Co Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ID-PRMD-1202
Record Dates: First submitted 2014-03-18; First posted 2014-04-04 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2013-04

CONDITIONS: Healthy
Keywords: Neuropathic pain; pregabalin
MeSH Terms: conditions — Neuralgia

ARMS (2):
- Immediate release capsule(lyrica capsule 150mg) (Active Comparator): Immediate release capsule repeat treatment for 3days under fasted condition
  Interventions: Drug: Immediate release capsule(lyrica 150mg * 2/day)
- sustained release tablet (Experimental): sustained release tablet repeat treatment for 3days under fasted condition
  Interventions: Drug: sustained release tablet

INTERVENTIONS:
Drug: Immediate release capsule(lyrica 150mg * 2/day) — Immediate release capsule
  Arms: Immediate release capsule(lyrica capsule 150mg)
Drug: sustained release tablet — sustained release tablet
  Arms: sustained release tablet

SUMMARY:
The purpose of this study is to compare the pharmacokinetics profiles of pregabalin sustained release tablet (300mg) to immediate release capsule(150mg * 2) while multiple dosing.

ELIGIBILITY:
Inclusion Criteria:

* 19~44 aged healthy adult.
* someone tho has at least 50kg body weight and ideal body weight ±20%

Exclusion Criteria:

* someone has acute symptom at screening phase
* someone has any disease or symptoms which is clinically significant
* someone had been determined during healthy examination in screening period
* AST or ALT > 1.25 times than normal
* Total bilirubin > 1.5 times than normal
* someone who has a history of allergy, anaphylaxis, drug abuse or misuse.
* someone who had enrolled to other clinical trial within the last 60 days.
* someone who had donated blood within the last 60 days.
* someone who can't take a meal derived from this trial.
* someone who has taken abnormal meals like which can affect to drug ADME
* someone who has taken other ETC drugs or oriental drugs within the last 14 days, Or OTC drugs within the last 7 days
* someone who has taken caffein continuously (coffee or green tea more than 5 cups per a day) or took caffein since 24hours before.
* someone who has taken alcohol more than 30g/day or smoked more than 10 piece of tobacco/day.
* someone who has galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption.

Ages: 19 Years to 44 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Measure blood concentration of pregabalin | 0~4day / 14~18day

SECONDARY OUTCOMES:
Safety evaluation | 0~25day

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic medical center, Seoul, Seocho-gu, South Korea